CLINICAL TRIAL: NCT07305883
Title: Intranasal Ketorolac Effectiveness In Comparison To Intranasal Ketamine for Digital Nerve Block Pain; A Randomized, Double Blind Trial
Brief Title: Comparison of Intranasal Ketorolac and Intranasal Ketamine in Digital Nerve Block Pain
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-5-243-91681
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pain; Digital Block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Ketamine (Active Comparator): 50 mg ketamine will be administered intranasally using mucosal atomizer,. Half dose (0.5cc) in each nostril, Given 5 minutes before digital nerve block
  Interventions: Drug: Intranasal ketamine
- Intranasal Ketorolac Tromethamine (Experimental): 30 mg ketorolac will be administered intranasally using mucosal atomizer. Half dose (0.5 cc) in each nostril, Given 5 minutes before digital nerve block.
  Interventions: Drug: Intranasal Ketorolac Tromethamine

INTERVENTIONS:
Drug: Intranasal Ketorolac Tromethamine — 30 mg ketorolac will be administered intranasally using mucosal atomizer. Half dose (0.5 cc) in each nostril, Given 5 minutes before digital nerve block.
  Arms: Intranasal Ketorolac Tromethamine
Drug: Intranasal ketamine — 50 mg ketamine will be administered intranasally using mucosal atomizer,. Half dose (0.5cc) in each nostril, Given 5 minutes before digital nerve block
  Arms: Intranasal Ketamine

SUMMARY:
This study aims to compare the analgesic effectiveness and side effects of intranasal ketorolac versus intranasal ketamine for reducing pain prior to digital nerve block procedures in patients with finger injuries in emergency department.

DETAILED DESCRIPTION:
Acute pain management in emergency department during painful procedures such as digital nerve block is crucial to be implemented in a rapid-onset method. Ketorolac, a potent NSAID, and ketamine, an NMDA receptor antagonist with analgesic effects, have both been shown to be effective and fast-onset when administered intranasally. This non-invasive method of Ketorolac is not supported by sufficient evidences in such clinical scenarios. Addressing this research gap may lead to reduced pain and complications, as well as higher patient satisfaction, contributing the development of novel pre-procedural analgesic strategies in emergency settings.

Participants will be randomly assigned to receive either 30 mg intranasal ketorolac or 50 mg intranasal ketamine, administered 5 minutes prior to the digital nerve block. Pain will be assessed using the Numeric Rating Scale (NRS). Secondary endpoints include nasal irritation, side effects, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Weight > 50 kg
* Requires digital nerve block
* Able to provide informed consent

Exclusion Criteria:

* Active peptic ulcer disease (PUD)
* History of hypersensitivity to NSAIDs
* Pregnancy and breastfeeding
* Renal failure
* Hepatic failure
* Patients who have received analgesics within the past 6 hours
* Nasal congestion
* Upper respiratory tract infection
* Patients with a history of kidney transplantation
* Active gastrointestinal bleeding
* Systolic blood pressure less than 90 mmHg or greater than 180 mmHg
* Heart rate less than 50 per minute or greater than 150 per minute
* Concurrent use of NSAIDs or anticoagulant drugs
* Inability to provide informed consent
* Anatomical abnormalities of the nose or skull base (congenital or acquired)
* Hyperreactive airway disease such as severe asthma
* Coagulation disorders
* Intracranial hemorrhage
* Suspected aortic dissection
* Suspected rupture of abdominal aortic aneurysm
* History of gastrointestinal perforation
* Gastrointestinal bleeding within the past month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Block pain intensity | Immediately after block
  The numerical rating score (NRS) will be used for the study. The NRS ranges from 0 (no pain) to 10 (very severe pain). The higher the pain scores the higher the pain severity. The pain severity will be asked from the patients.

SECONDARY OUTCOMES:
Nasal irritation | 60 minutes after the block
  We will ask the patients about this outcome use a 3-level Likert-like scale.
Side effects | From the drug administration to 60 minutes after the block
  The patients will be assessed every 15 minutes for this outcome.
Patient satisfaction score | 60 minutes after the drug administration.
  The patients will be asked about their satisfaction using a 3-level Likert like scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Mirfazaelian, Principal Investigator — Tehran University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No
The information is not allowed to be shared.